CLINICAL TRIAL: NCT05478356
Title: The Effects of Low-dose Atropine and Orthokeratology in Pediatric Myopia Control
Acronym: AVO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Evidence Based Cataract Study Group (Other)
Responsible Party: Principal Investigator, Peng ZHOU, Doctor, Evidence Based Cataract Study Group
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EvidenceBCSG
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- orthokeratology group (Experimental)
  Interventions: Device: orthokeratology
- low-dose atropine group (Active Comparator)
  Interventions: Drug: low-dose atropine eye drops

INTERVENTIONS:
Drug: low-dose atropine eye drops — low-dose atropine eye drops
  Arms: low-dose atropine group
Device: orthokeratology — orthokeratology, ortho-K lenses
  Arms: orthokeratology group

SUMMARY:
Both orthokeratology and atropine eye drops are effective methods for myopia control, but few studies have compared them all together simultaneously. Therefore, the primary aim of the present study was to compare the effect of orthokeratology versus low-dose (0.01% and 0.02%) atropine on the control of myopia progression.

ELIGIBILITY:
Inclusion Criteria:

Best corrected visual acuity less then 0.00 log MAR (minimum angle of resolution) units Cycloplegic SER of - 1.0 D or less in both eyes. An inter-eye cycloplegic SER difference of 1.00 D or more.

Exclusion Criteria:

Children with cycloplegic cylinder refraction of more than + 1.00 D or less than - 1.00 D.

History of binocular vision problems, including strabismus. History of known ocular disorders, including media opacities, macular dysgenesis, optic nerve hypoplasia, perinatal brain injury, buphthalmos, and retinopathy of prematurity.

History of medication use that might have affected the refractive results. Systemic or developmental problems that might have hindered refractive development.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression of myopia | 1 year
  The change of myopia (Ds)
Progression of axial length | 1 year
  The change of axial length (mm)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Visionly Eye Hospital, Beijing, Beijing Municipality
  - Parkway Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided